CLINICAL TRIAL: NCT01246063
Title: A Phase I/II Trial of Carfilzomib, Pegylated Liposomal Doxorubicin, and Dexamethasone for the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: Carfilzomib, Pegylated Liposomal Doxorubicin Hydrochloride, and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201102043
Record Dates: First submitted 2010-11-15; First posted 2010-11-23 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; liposomal doxorubicin; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase I - Part 1 Dose Level 0 (Carfilzomib 20/27 mg/m^2) (Experimental): Dose Level 0: Carfilzomib IV (20 mg/m^2) D1&D2 of C1 and carfilzomib IV (27 mg/m^2)D8, D9, D15, D16 of C1. Carfilzomib IV (27 mg/m^2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (27 mg/m^2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m^2)D8 C1-6.
  Interventions: Drug: carfilzomib; Drug: pegylated liposomal doxorubicin (PLD)
- Phase I - Part 1 Dose Level 1 (Carfilzomib 20/36 mg/m^2) (Experimental): Dose Level 1: Carfilzomib IV (20 mg/m^2) D1&D2 of C1 and carfilzomib IV (36 mg/m^2)D8, D9, D15, D16 of C1. Carfilzomib IV (36 mg/m^2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (36 mg/m^2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m^2)D8 C1-6.
  Dose Level 1: Carfilzomib IV (1 dose level above MTD) D1, D2, D8, D9, D15, D16 C1-6. Carfilzomib IV (1 dose level above MTD) D1, D8, D15, D22 C7 and subsequent cycles. PLD IV (1 dose level above MTD) D8 of each cycle. Dexamethasone 20 mg IV or PO same schedule as carfilzomib.
  Dose Level 2: Carfilzomib IV (2 dose levels above MTD) D1, D2, D8, D9, D15, D16 C1-6. Carfilzomib IV (2 dose levels above MTD) D1, D8, D15, D22 C7 and subsequent cycles. PLD IV (2 dose levels above MTD) D8 of each cycle. Dexamethasone 20 mg IV or PO same schedule as carfilzomib.
  Interventions: Drug: carfilzomib; Drug: pegylated liposomal doxorubicin (PLD)
- Phase I - Part 1 Dose Level 2 (Carfilzomib 20/45 mg/m^2) (Experimental): Dose Level 2: Carfilzomib IV (20 mg/m^2) D1&D2 of C1 and carfilzomib IV (45 mg/m^2)D8, D9, D15, D16 of C1. Carfilzomib IV (45 mg/m^2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (45 mg/m^2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m^2)D8 C1-6.
  Interventions: Drug: carfilzomib; Drug: pegylated liposomal doxorubicin (PLD)
- Phase I - Part 1 Dose Level 3 (Carfilzomib 20/56 mg/^2) (Experimental): Dose Level 3: Carfilzomib IV (20 mg/m^2) D1&D2 of C1 and carfilzomib IV (56 mg/m^2)D8, D9, D15, D16 of C1. Carfilzomib IV (56 mg/m^2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (56 mg/m^2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m^2)D8 C1-6.
  Interventions: Drug: carfilzomib; Drug: pegylated liposomal doxorubicin (PLD)
- Phase I -Part 2 Cohort 0 (Carfilzomib 56 mg/m^2+Dexamethasone) (Experimental): Cohort 0: Carfilzomib IV (56 mg/^2 - Phase 1 Part 1) D1, D2, D8, D9, D15, D16 C1-6. Carfilzomib IV (56 mg/m^2 - Phase 1 Part 1) D1, D8, D15, D22 C7 and subsequent cycles. PLD IV (30 mg/m^2 - Phase 1 Part 1) D8 of each cycle. Dexamethasone 20 mg IV or PO same schedule as carfilzomib.
  Interventions: Drug: carfilzomib; Drug: pegylated liposomal doxorubicin (PLD); Drug: Dexamethasone
- Phase 2 (Carfilzomib 56 mg/m^2+ Dexamethasone) (Experimental): Carfilzomib IV (56 mg/^2 - Phase 1 Part 1) D1, D2, D8, D9, D15, D16 C1-6. Carfilzomib IV (56 mg/m^2 - Phase 1 Part 1) D1, D8, D15, D22 C7 and subsequent cycles. PLD IV (30 mg/m^2 - Phase 1 Part 1) D8 of each cycle. Dexamethasone 20 mg IV or PO same schedule as carfilzomib.
  Interventions: Drug: carfilzomib; Drug: pegylated liposomal doxorubicin (PLD); Drug: Dexamethasone

INTERVENTIONS:
Drug: carfilzomib
  Other Names: Kyprolis; CFZ
Drug: pegylated liposomal doxorubicin (PLD)
  Other Names: DOXIL
Drug: Dexamethasone
  Other Names: Decadron
  Arms: Phase 2 (Carfilzomib 56 mg/m^2+ Dexamethasone); Phase I -Part 2 Cohort 0 (Carfilzomib 56 mg/m^2+Dexamethasone)

SUMMARY:
The aim of this phase I/II trial is to determine the maximal tolerated dose (MTD) of carfilzomib together with pegylated liposomal doxorubicin hydrochloride (PLD) with or without dexamethasone, and then to establish the efficacy and safety of this novel combination in patients with relapsed or refractory multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of multiple myeloma with a measurable disease parameter at time of screening; a measurable disease parameter is defined as one or more of the following:

  * Serum monoclonal protein >= 0.5 g/dl
  * 24 hour urine monoclonal protein >= 0.2 g/24 hour
  * Serum free light chain ratio > 5 x normal ratio with an absolute difference of 10mg/dl between the involved and uninvolved free light chain
  * Soft tissue plasmacytoma >= 2 cm measurable by either physical examination and/or applicable radiographs (e.g. magnetic resonance imaging [MRI], computed tomography [CT], etc)
  * Bone Marrow Plasma Cells >= 30%
* Documentation of at least one line of prior myeloma therapy now with relapsed or refractory disease requiring re-treatment
* At least 18 years of age at the time of signing the informed consent.
* Performance status of Eastern Cooperative Oncology Group (ECOG) =< 2 or Karnofsky >= 60%; participants with lower performance status based solely on bone pain secondary to multiple myeloma will be eligible
* Required laboratory values

  * Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) and aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) < 2.5 x the upper limit of the institutional normal value (ULN)
  * Total bilirubin =< 1.5 x upper limit of normal (ULN)
  * Absolute neutrophil count (ANC) >= 1,000
  * Hemoglobin >= 8 g/dl
  * Platelets >= 50,000
  * Creatinine clearance > 15 ml/minute using Cockcroft-Gault formula
  * For those participants receiving warfarin (Coumadin), unfractionated heparin, or low-molecular weight heparin therapy, the applicable coagulation parameter that is being monitored must be within the accepted therapeutic ranges for those indications
  * Transfusions and/or growth factor dependent participants are not excluded if the above parameters can be achieved with such support
* Females of childbearing potential (FCBP) must agree to refrain from becoming pregnant while on study drug and for 3 months after discontinuation from study drug, and must agree to use adequate contraception including hormonal contraception, (i.e. birth control pills, etc), barrier method contraception (i.e. condoms), or abstinence during that time frame; FCBP must agree to regular pregnancy testing during this timeframe; inclusion of FCBP requires two negative pregnancy tests prior to enrollment. All women, regardless of age, should be considered FCBP unless they are surgically sterile (post hysterectomy, post bilateral oophorectomy, etc) or have been naturally post menopausal for >= 24 consecutive months
* Men engaging in sexual intercourse with a FCBP must agree to use adequate contraception including hormonal contraception, (i.e. birth control pills, etc), barrier method contraception (i.e. condoms), or abstinence while on study drug and for 3 months after discontinuation from study drug
* Ability to understand and willing to sign a written informed consent document

Exclusion Criteria:

* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Plasma Cell Leukemia
* Waldenstrom's macroglobulinemia
* Pregnant or lactating females
* Use of any anti-myeloma drug therapy within 14 days of initiation of study drug treatment excluding corticosteroids if given for an indication other than myeloma; bisphosphonates are not considered anti-myeloma drugs
* Participation in an investigational therapeutic study within 14 days of initiation of study drug treatment
* Radiotherapy to multiple sites or immunotherapy within 14 days of initiation of study drug treatment (localized radiotherapy to a single site at least 7 days before start is permissible)
* Major surgery within 14 days of initiation of study drug treatment
* Participants in whom the required program of oral (PO) and IV fluid hydration is contraindicated
* Prior history of a hypersensitivity reaction to PLD, doxorubicin, bortezomib, carfilzomib, or liposomal drug formulations other than PLD; history of reactions to liposomal drug formulations other than PLD should be evaluated individually and if their reactions were felt to have been due to the encapsulated agent, rather than the liposomal component itself they should be excluded at the discretion of the investigators
* Participants who are known to have active hepatitis A, B, or C viral infection may not participate in this study; active disease is defined as participants with a known viral hepatitis whose liver function tests are elevated
* Known human immunodeficiency virus (HIV)-seropositive and are taking anti-retrovirals may not participate in this study; participants who are HIV-seropositive and not on anti-retroviral therapy and who otherwise meet the inclusion/exclusion criteria will be eligible for the study
* Compromised cardiovascular function defined as any of the following:

  * Electrocardiogram (EKG) evidence of acute ischemia
  * EKG evidence of medically significant conduction system abnormalities
  * History of myocardial infarction within the last 6 months
  * Unstable angina pectoris or cardiac arrhythmia
  * History of Class 3 or Class 4 New York Heart Association Congestive Heart Failure within 6 months of enrollment on study
  * Left ventricular ejection fraction (LVEF) < 45% by either echocardiography or radionuclide-based multiple gated acquisition (Echo or MUGA)
* Uncontrolled concurrent illness including: other hematologic or non-hematologic malignancy, active infection, or uncontrolled diabetes
* Any significant psychological, medical, or surgical condition thought to compromise the participant, the study, or prevent informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05-14 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2018-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schroeder MA, Fiala MA, Huselton E, Cardone MH, Jaeger S, Jean SR, Shea K, Ghobadi A, Wildes T, Stockerl-Goldstein KE, Vij R. A Phase I/II Trial of Carfilzomib, Pegylated Liposomal Doxorubicin, and Dexamethasone for the Treatment of Relapsed/Refractory Multiple Myeloma. Clin Cancer Res. 2019 Jul 1;25(13):3776-3783. doi: 10.1158/1078-0432.CCR-18-1909. Epub 2019 Apr 5. PMID 30952640
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 05/14/2012 and closed to participant enrollment on 08/02/2016.
Groups:
- Phase I - Part 1 Dose Level 1 (Carfilzomib 20/36 mg/m^2): Dose Level 1: Carfilzomib IV (20 mg/m^2) D1&D2 of C1 and carfilzomib IV (36 mg/m^2)D8, D9, D15, D16 of C1. Carfilzomib IV (36 mg/m^2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (36 mg/m^2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m^2)D8 C1-6.
Period: Overall Study
Arm/Group | Phase I - Part 1 Dose Level 0 (Carfilzomib 20/27 mg/m^2) | Phase I - Part 1 Dose Level 1 (Carfilzomib 20/36 mg/m^2) | Phase I - Part 1 Dose Level 2 (Carfilzomib 20/45 mg/m^2) | Phase I - Part 1 Dose Level 3 (Carfilzomib 20/56 mg/^2) | Phase I -Part 2 Cohort 0 (Carfilzomib 56 mg/m^2+Dexamethasone) | Phase 2 (Carfilzomib 56 mg/m^2+ Dexamethasone)
Started | 3 | 4 | 4 | 5 | 7 | 17
Completed | 3 | 4 | 4 | 5 | 7 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I - Part 1 Dose Level 0 (Carfilzomib 20/27 mg/m^2): Dose Level 0: Carfilzomib IV (20 mg/m2) D1&D2 of C1 and carfilzomib IV (27 mg/m2)D8, D9, D15, D16 of C1. Carfilzomib IV (27 mg/m2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (27 mg/m2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m2)D8 C1-6.
- Phase I - Part 1 Dose Level 1 (Carfilzomib 20/36 mg/m^2): Dose Level 1: Carfilzomib IV (20 mg/m2) D1&D2 of C1 and carfilzomib IV (36 mg/m2)D8, D9, D15, D16 of C1. Carfilzomib IV (36 mg/m2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (36 mg/m2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m2)D8 C1-6.
- Phase I - Part 1 Dose Level 2 (Carfilzomib 20/45 mg/m^2): Dose Level 2: Carfilzomib IV (20 mg/m2) D1&D2 of C1 and carfilzomib IV (45 mg/m2)D8, D9, D15, D16 of C1. Carfilzomib IV (45 mg/m2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (45 mg/m2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m2)D8 C1-6.
- Phase I - Part 1 Dose Level 3 (Carfilzomib 20/56 mg/^2): Dose Level 3: Carfilzomib IV (20 mg/m2) D1&D2 of C1 and carfilzomib IV (56 mg/m2)D8, D9, D15, D16 of C1. Carfilzomib IV (56 mg/m2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (56 mg/m2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m2)D8 C1-6.
- Phase I-Part 2 Cohort 0 (Carfilzomib 56 mg/m^2+Dexamethasone): Cohort 0: Carfilzomib IV (56 mg/^2 - Phase 1 Part 1) D1, D2, D8, D9, D15, D16 C1-6. Carfilzomib IV (56 mg/m^2 - Phase 1 Part 1) D1, D8, D15, D22 C7 and subsequent cycles. PLD IV (30 mg/m^2 - Phase 1 Part 1) D8 of each cycle. Dexamethasone 20 mg IV or PO same schedule as carfilzomib.
- Total: Total of all reporting groups
Arm/Group | Phase I - Part 1 Dose Level 0 (Carfilzomib 20/27 mg/m^2) | Phase I - Part 1 Dose Level 1 (Carfilzomib 20/36 mg/m^2) | Phase I - Part 1 Dose Level 2 (Carfilzomib 20/45 mg/m^2) | Phase I - Part 1 Dose Level 3 (Carfilzomib 20/56 mg/^2) | Phase I-Part 2 Cohort 0 (Carfilzomib 56 mg/m^2+Dexamethasone) | Phase 2 (Carfilzomib 56 mg/m^2+ Dexamethasone) | Total
Number analyzed (Participants) | 3 | 4 | 4 | 5 | 7 | 17 | 40
Age, Continuous [Median (Full Range); unit: years] | 65 [62 to 66] | 66.5 [53 to 71] | 72 [55 to 79] | 57 [54 to 69] | 63 [27 to 67] | 65 [46 to 70] | 65 [27 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 5 | 5 | 7 | 23
  Male | 1 | 2 | 2 | 0 | 2 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 4 | 4 | 4 | 7 | 17 | 37
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 0 | 5 | 9
  White | 2 | 3 | 3 | 4 | 7 | 11 | 30
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 4 | 4 | 5 | 7 | 17 | 40

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Carfilzomib and Pegylated Liposomal Doxorubicin (Phase I - Part 1).
Description: * MTD is the maximum tolerated dose level tested unless dose limiting toxicity (DLT) are observed during Cycle 1. If DLT is observed, MTD will be the next lower dose level.
  * Please note that the maximum tolerated dose of carfilzomib and pegylated liposomal doxorubicin was not reached. The data below is the recommended dosage for further studies.
Time Frame: 28 days (completion of first cycle of all Phase I - Part 1 patients)
Population: Participants enrolled in the Phase I - Part 1 portion of this study were the only evaluable participants for this outcome measure.
Measure: Number; unit: mg/m^2
Groups:
- Phase I - Part 1: Dose Level 0: Carfilzomib IV (20 mg/m^2) D1&D2 of C1 and carfilzomib IV (27 mg/m^2)D8, D9, D15, D16 of C1. Carfilzomib IV (27 mg/m^2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (27 mg/m^2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m^2)D8 C1-6.
  Dose Level 1: Carfilzomib IV (20 mg/m^2) D1&D2 of C1 and carfilzomib IV (36 mg/m^2)D8, D9, D15, D16 of C1. Carfilzomib IV (36 mg/m^2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (36 mg/m^2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m^2)D8 C1-6.
  Dose Level 2: Carfilzomib IV (20 mg/m^2) D1&D2 of C1 and carfilzomib IV (45 mg/m^2)D8, D9, D15, D16 of C1. Carfilzomib IV (45 mg/m^2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (45 mg/m^2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m^2)D8 C1-6.
  Dose Level 3: Carfilzomib IV (20 mg/m^2) D1&D2 of C1 and carfilzomib IV (56 mg/m^2)D8, D9, D15, D16 of C1. Carfilzomib IV (56 mg/m^2) D1, D2, D8, D9, D15, D16 C2-6. Carfilzomib IV (56 mg/m^2)D1, D2, D8, D15, D22 C7+. PLD IV (30 mg/m^2)D8 C1-6.
- Phase I - Part 2: Cohort 0: Carfilzomib IV (56 mg/^2 - Phase 1 Part 1) D1, D2, D8, D9, D15, D16 C1-6. Carfilzomib IV (56 mg/m^2 - Phase 1 Part 1) D1, D8, D15, D22 C7 and subsequent cycles. PLD IV (30 mg/m^2 - Phase 1 Part 1) D8 of each cycle. Dexamethasone 20 mg IV or PO same schedule as carfilzomib.
- Phase 2: Carfilzomib IV (56 mg/^2 - Phase 1 Part 1) D1, D2, D8, D9, D15, D16 C1-6. Carfilzomib IV (56 mg/m^2 - Phase 1 Part 1) D1, D8, D15, D22 C7 and subsequent cycles. PLD IV (30 mg/m^2 - Phase 1 Part 1) D8 of each cycle. Dexamethasone 20 mg IV or PO same schedule as carfilzomib.
Arm/Group | Phase I - Part 1 | Phase I - Part 2 | Phase 2
Number analyzed (Participants) | 16 | 0 | 0
mg/m^2
  Carfilzomib Recommended Dose | 56 |  |
  Pegylated liposomal doxorubicin recommended dose | 30 |  |

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Carfilzomib and PLD (Phase I - Part 2).
Description: -MTD is the maximum tolerated dose level tested unless dose limiting toxicity (DLT) are observed during Cycle 1. If DLT is observed, MTD will be the next lower dose level.
Time Frame: 28 days (completion of first cycle of all Phase I - Part 2 patients)
Population: Participants enrolled in the Phase I - Part 2 portion of this study were the only evaluable participants for this outcome measure.
Measure: Number; unit: mg/m^2
Arm/Group | Phase I - Part 1 | Phase I - Part 2 | Phase 2
Number analyzed (Participants) | 0 | 7 | 0
mg/m^2
  Carfilzomib dose |  | 56 |
  Pegylated liposomal doxorubicin dose |  | 30 |

3. Primary Outcome: Maximum Tolerated Dose (MTD) of Dexamethasone (Phase I - Part 2).
Description: as for outcome 2
Time Frame: 28 days (completion of first cycle of all Phase I - Part 2 patients)
Population: as for outcome 2
Measure: Number; unit: mg
Arm/Group | Phase I - Part 1 | Phase I - Part 2 | Phase 2
Number analyzed (Participants) | 0 | 7 | 0
mg |  | 20 |

4. Primary Outcome: Phase 2 - Efficacy of Carfilzomib in Combination With PLD and Dexamethasone as Measured by the Percentage of Participants With Confirmed Tumor Responses
Description: -A confirmed response is defined to be a complete response (CR), very good partial response (VGPR), or partial response (PR) per IMWG Criteria.
Time Frame: Completion of treatment (median number of cycles was 9.5 (range 1-34))
Population: For this outcome measure the Phase I - Part 1 Dose Level 3 and Phase I - Part 2 participants were combined with the Phase 2 participants as they received the same dosing of carfilzomib. The remaining Phase I - Part 1 participants were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 (Includes Phase I - Part 2 Participants): Phase I Part 2 Cohort 0: Carfilzomib IV (56 mg/^2 - Phase 1 Part 1) D1, D2, D8, D9, D15, D16 C1-6. Carfilzomib IV (56 mg/m^2 - Phase 1 Part 1) D1, D8, D15, D22 C7 and subsequent cycles. PLD IV (30 mg/m^2 - Phase 1 Part 1) D8 of each cycle. Dexamethasone 20 mg IV or PO same schedule as carfilzomib.
  Phase 2: Carfilzomib IV (56 mg/^2 - Phase 1 Part 1) D1, D2, D8, D9, D15, D16 C1-6. Carfilzomib IV (56 mg/m^2 - Phase 1 Part 1) D1, D8, D15, D22 C7 and subsequent cycles. PLD IV (30 mg/m^2 - Phase 1 Part 1) D8 of each cycle. Dexamethasone 20 mg IV or PO same schedule as carfilzomib.
Arm/Group | Phase I - Part 1 | Phase 2 (Includes Phase I - Part 2 Participants)
Number analyzed (Participants) | 0 | 24
Participants |  | 20

5. Primary Outcome: Phase 2 - Toxicity of Carfilzomib in Combination With PLD and Dexamethasone as Measured by Number of Participants Who Experience Grade 3/4 Toxicity
Time Frame: Through 30 days after completion of treatment (median number of cycles was 9.5 (range 1-34))
Population: For this outcome measure the Phase I - Part 2 participants were combined with the Phase 2 participants as they received the same dosing regimen. Phase I - Part 1 participants were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Part 1 | Phase 2 (Includes Phase I - Part 2 Participants)
Number analyzed (Participants) | 0 | 24
Participants |  | 22

6. Secondary Outcome: Median Overall Survival
Time Frame: Completion of follow-up (median of 23.3 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I - Part 1 Dose Level 0 (Carfilzomib 20/27 mg/m^2) | Phase I - Part 1 Dose Level 1 (Carfilzomib 20/36 mg/m^2) | Phase I - Part 1 Dose Level 2 (Carfilzomib 20/45 mg/m^2) | Phase I - Part 1 Dose Level 3 (Carfilzomib 20/56 mg/^2) | Phase I-Part 2 Cohort 0 (Carfilzomib 56 mg/m^2+Dexamethasone) | Phase 2 (Carfilzomib 56 mg/m^2+ Dexamethasone)
Number analyzed (Participants) | 3 | 4 | 4 | 5 | 7 | 17
months | 25.490 [.000 to 60.025] | 18.780 [1.493 to 36.067] | 11.610 [.000 to 23.889] | 32.340 [.000 to 86.811] | 18.720 [8.660 to 28.780] | NA [NA to NA] — The median overall survival was not reached in the follow-up time period.

7. Secondary Outcome: Progression-free Survival Time (Phase 2 Only)
Description: -Progression per IMWG Criteria
Time Frame: Through completion of follow-up (median follow-up was 23.3 months)
Population: This outcome measure is for Phase 2 (including Phase I Part 2) participants only. Phase I Part 2 and Phase 2 participants who began alternative anti-multiple myeloma treatment prior to progression were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I - Part 1 | Phase 2 (Includes Phase I - Part 2 Participants)
Number analyzed (Participants) | 0 | 8
months |  | 13.4 [5.0 to 21.7]

8. Secondary Outcome: Median Duration of Overall Response
Description: * For participants with confirmed tumor responses
  * A confirmed response is defined to be a complete response (CR), very good partial response (VGPR), or partial response (PR) per IMWG Criteria
Time Frame: Through completion of follow-up (median follow-up was 23.3 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I - Part 1 Dose Level 0 (Carfilzomib 20/27 mg/m^2) | Phase I - Part 1 Dose Level 1 (Carfilzomib 20/36 mg/m^2) | Phase I - Part 1 Dose Level 2 (Carfilzomib 20/45 mg/m^2) | Phase I - Part 1 Dose Level 3 (Carfilzomib 20/56 mg/^2) | Phase I-Part 2 Cohort 0 (Carfilzomib 56 mg/m^2+Dexamethasone) | Phase 2 (Carfilzomib 56 mg/m^2+ Dexamethasone)
Number analyzed (Participants) | 1 | 2 | 2 | 4 | 5 | 15
months | 6.090 [NA to NA] — The 95% confidence interval was not estimable as no one was censored so the numbers are actuals and not estimates. | 6.840 [NA to NA] — The 95% confidence interval was not estimable as no one was censored so the numbers are actuals and not estimates. | 3.420 [NA to NA] — The 95% confidence interval was not estimable as no one was censored so the numbers are actuals and not estimates. | 13.130 [.000 to 27.761] | 9.440 [3.580 to 15.300] | 23.950 [14.072 to 33.828]

ADVERSE EVENTS:
Time Frame: Adverse events were followed from first day of study treatment until 30 days following the last day of study treatment or until the start of a new chemotherapy, whichever is sooner. Median number of cycles was 9.5 (range 1-34 cycles). All-cause mortality data was collected from first day of study treatment until completion of treatment.
Arm/Group | Phase I - Part 1 Dose Level 0 (Carfilzomib 20/27 mg/m^2) | Phase I - Part 1 Dose Level 1 (Carfilzomib 20/36 mg/m^2) | Phase I - Part 1 Dose Level 2 (Carfilzomib 20/45 mg/m^2) | Phase I - Part 1 Dose Level 3 (Carfilzomib 20/56 mg/^2) | Phase I -Part 2 Cohort 0 (Carfilzomib 56 mg/m^2+Dexamethasone) | Phase 2 (Carfilzomib 56 mg/m^2+ Dexamethasone)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 2/4 | 0/5 | 0/7 | 1/17
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/4 | 4/4 | 3/5 | 2/7 | 10/17
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 4/4 | 5/5 | 7/7 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Part 1 Dose Level 0 (Carfilzomib 20/27 mg/m^2) (N=3) | Phase I - Part 1 Dose Level 1 (Carfilzomib 20/36 mg/m^2) (N=4) | Phase I - Part 1 Dose Level 2 (Carfilzomib 20/45 mg/m^2) (N=4) | Phase I - Part 1 Dose Level 3 (Carfilzomib 20/56 mg/^2) (N=5) | Phase I -Part 2 Cohort 0 (Carfilzomib 56 mg/m^2+Dexamethasone) (N=7) | Phase 2 (Carfilzomib 56 mg/m^2+ Dexamethasone) (N=17)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aortic valve disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
Infusion related reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Weakness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
RSV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 1
Skin infection (cellulitis) (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (MRSA) (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (shingles) (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Polypharmacy (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Left hip pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Acute encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute rental failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnea (COPD exacerbation) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thromboembolic event (DVT) (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Part 1 Dose Level 0 (Carfilzomib 20/27 mg/m^2) (N=3) | Phase I - Part 1 Dose Level 1 (Carfilzomib 20/36 mg/m^2) (N=4) | Phase I - Part 1 Dose Level 2 (Carfilzomib 20/45 mg/m^2) (N=4) | Phase I - Part 1 Dose Level 3 (Carfilzomib 20/56 mg/^2) (N=5) | Phase I -Part 2 Cohort 0 (Carfilzomib 56 mg/m^2+Dexamethasone) (N=7) | Phase 2 (Carfilzomib 56 mg/m^2+ Dexamethasone) (N=17)
Anemia (Blood and lymphatic system disorders) | 0 | 3 | 4 | 4 | 6 | 14
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 2
Lymph node swelling (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Heart murmur (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 1
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 2 | 2
Right ear fullness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Blurred vision (Eye disorders) | 0 | 0 | 2 | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 4
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eye erythema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flashing lights (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Subconjunctival hemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Watering eyes (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 3 | 2 | 1 | 6
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 3 | 5 | 4 | 9
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypersalivating (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Indigestion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mouth sores (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mucositits oral (Gastrointestinal disorders) | 0 | 0 | 2 | 4 | 1 | 6
Nausea (Gastrointestinal disorders) | 3 | 1 | 3 | 4 | 4 | 9
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sores at corner of mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Stomach flu (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomach virus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Upset stomach (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 2 | 2 | 6 | 4
Achy (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Black spot-tongue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 2 | 4 | 1 | 4
Edema face (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Edema limbs (General disorders) | 2 | 1 | 1 | 1 | 0 | 2
Fatigue (General disorders) | 3 | 2 | 3 | 5 | 5 | 10
Fever (General disorders) | 1 | 0 | 3 | 4 | 2 | 8
Flu Like Symptoms (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Generalized pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 3
Groin pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hand pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
IV site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 2 | 5
Injection like reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Kidney pain cramping (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Legs/jaw/head pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 0 | 1 | 1 | 5
Localized edema-feet (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 2 | 0 | 2
Neck edema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (General disorders) | 0 | 0 | 0 | 1 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 2
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rib cage pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Shoulder blade pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sweating (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Gallstones (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bone infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
C. diff colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Finger wart (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Groin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Oral candidiasis/thrush (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 5
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pain-head to toe (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Perianal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Salivary gland infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 3 | 2 | 5
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Stool (+) VRE (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Stool (+) norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Stye (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 2 | 0 | 2 | 4 | 3 | 10
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 4
Viral illness (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Elbow wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 2 | 0 | 3
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Great toe wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Phalangeal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Rib fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Right foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Spinal fracture - pathologic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 3 | 3 | 3 | 10
Alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 1 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 3 | 3 | 4 | 14
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 2 | 2 | 5
CPK increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Cardiac troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Cholesterol high (Investigations) | 0 | 0 | 0 | 1 | 0 | 3
Creatinine increased (Investigations) | 3 | 2 | 3 | 3 | 5 | 8
INR increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 6
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 3 | 1 | 3 | 4 | 7 | 17
Lymphocyte count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 1 | 4 | 6 | 12
Platelet count decreased (Investigations) | 2 | 1 | 3 | 5 | 7 | 17
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Weight gain (Investigations) | 0 | 0 | 0 | 1 | 2 | 1
Weight loss (Investigations) | 0 | 1 | 0 | 3 | 0 | 5
White blood cell decreased (Investigations) | 1 | 2 | 3 | 3 | 5 | 17
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 4 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 3 | 6
Diabetes type 2 (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 3 | 9
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 7
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 3
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 1 | 8
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 5 | 12
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 3 | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 2 | 4 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 3 | 4 | 5 | 5 | 6
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 4 | 4 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 4 | 1 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 2 | 3 | 12
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Achiness hips (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2 | 1 | 2
Body aches (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 1 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cramping arms, hands, and feet (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cramping hands and feet (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Elbow pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2
Foot pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3
Hip/leg pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intercostal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Joint range of motion decreased in lumbar spine (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Muscle cramps/spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms-hands (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle weakness-hands (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle weakness/heaviness lower limbs (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Osteonecrosis of palate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Rib pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2
Right armpit pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Right rib cage pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Right side pain with deep breath (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rotator cuff tear full/partial (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2
Shoulder spasm (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Warm spot on thigh (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Wrist pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
BCCA Nasal Ala (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Enlarging pulmonary nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
T10 lesion-invasion into spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 2 | 5
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0
Facial droop (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Fingertip sensitivity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 3 | 4 | 8
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia-shingles pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 2 | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1 | 0 | 0 | 2 | 3
Sinus pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 2
Tingling/numbness lower jaw (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2 | 3
Concentration impairment (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1 | 3 | 2 | 1 | 4
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 3 | 9
ATN (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 1 | 0
Congestion head/chest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 4 | 3 | 10
Dypnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 3 | 4 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Indeterminate lung nodules (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 3 | 9
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Respiratory distress-tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 1 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
"Pink Areas" palms of hands (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Blood blisters (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Bug bites (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cat bite (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 3
Enlarging mole (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythematous rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flaking skin on hands (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Foot blisters (after excessive walking) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Head nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Open area-left eyebrow (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 0 | 2
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Petechial rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Poison ivy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1
Pressure ulcers - buttocks (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 1
Rash aceniform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash arms (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash-back (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin blisters s/p lesion removal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin tear (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Swelling from bug bites (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colonoscopy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Cytoscopy with bladder biopsies (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0
Excision osteonecrosis-maxilla (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Foot surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Shoulder rotator cuff repair-right (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Urethral sling placement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 1
Flushing-face (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 1
Hypertension (Vascular disorders) | 2 | 0 | 1 | 3 | 1 | 6
Hypotension (Vascular disorders) | 0 | 0 | 2 | 2 | 0 | 3
Thromboembolic event - DVT (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT01246063/Prot_SAP_ICF_000.pdf